CLINICAL TRIAL: NCT04690777
Title: Efficacy of Vestibular Physiotherapy Against Multi-component Exercise in Functional Improvement in the Elderly": Pilot Study of a Randomized Clinical Trial
Brief Title: Efficacy of Vestibular Physiotherapy Against Multi-component Exercise in Functional Improvement in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, MARINA LOPEZ GARCIA, Associate Professor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2410-N-19
Record Dates: First submitted 2020-12-19; First posted 2020-12-31 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Physical Therapy; Sports Physical Therapy; Exercise Therapy; Gait

STUDY DESIGN:
Intervention Model Description: This pilot study is a controlled and randomized clinical trial (simple ER) with two groups in parallel, comparing the combination of a multi-component therapeutic exercise protocol (MS) versus vestibular exercises (EVs) in over 70 years. participants were randomly assigned to the therapeutic exercise group or the vestibular exercise group
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VESTIBULAR EXERCISE at home telerehabilitation (Experimental): 1. The vestibular exercises were performed with the indications of a physical therapist, in sessions of about 20 minutes with 5 times per week (Monday to Friday) consisting of 5 repetitions ensuring the following were not overworked:
  1. Head and eye movements while sitting.
  2. Head and body movements while sitting.
  3. Paused exercises.
  4. Combined exercises of modifications on rungs, unstable surfaces and walking exercises.
  Interventions: Procedure: Experimental: VESTIBULAR EXERCISE
- MULTICOMPONENT EXERCISE at home telerehabilitaion (Experimental): 1. A 6-week multi-component therapeutic physical exercise program was carried out. The ministerial guide and the "Vivifrail" consensus was followed (25, 26). There were 5 daily sessions per week (Monday to Friday), each lasting approximately 45 minutes. These sessions were conducted following the instructions of a physical therapist. VIVIFRAIL exercises are intended to be used over a progression period of up to 12 weeks, with combined exercises by days in cardiovascular aerobic balance strength and flexibility.
  Interventions: Procedure: MULTICOMPONENT EXERCISE
- VESTIBULAR EXERCISE in clinic (Experimental): 1. The vestibular exercises were performed with the indications of a physical therapist, in sessions of about 20 minutes with 5 times per week (Monday to Friday) consisting of 5 repetitions ensuring the following were not overworked:
  1. Head and eye movements while sitting.
  2. Head and body movements while sitting.
  3. Paused exercises.
  4. Combined exercises of modifications on rungs, unstable surfaces and walking exercises.
  Interventions: Procedure: Experimental: VESTIBULAR EXERCISE
- multi component exercise in clinic (Experimental): 1. A 6-week multi-component therapeutic physical exercise program was carried out. The ministerial guide and the "Vivifrail" consensus was followed (25, 26). There were 5 daily sessions per week (Monday to Friday), each lasting approximately 45 minutes. These sessions were conducted following the instructions of a physical therapist. VIVIFRAIL exercises are intended to be used over a progression period of up to 12 weeks, with combined exercises by days in cardiovascular aerobic balance strength and flexibility.
  Interventions: Procedure: MULTICOMPONENT EXERCISE

INTERVENTIONS:
Procedure: Experimental: VESTIBULAR EXERCISE — OCULAR AND MOVEMENT EXERCISES
  Arms: VESTIBULAR EXERCISE at home telerehabilitation; VESTIBULAR EXERCISE in clinic
Procedure: MULTICOMPONENT EXERCISE — exercises includes strengthening, cardiovascular training, flexibility and balance
  Arms: MULTICOMPONENT EXERCISE at home telerehabilitaion; multi component exercise in clinic

SUMMARY:
Loss of vestibular function occurs normally with healthy aging but can produce symptoms that reduce motor skills and cause falls. vestibular physical therapy (VPH) exercises are a specific approach to reducing imbalances. The multicomponent therapeutic physical exercise (ME) is an effective non-pharmacological strategy for the improvement of physical condition.

Objective: to determine the efficacy of ME versus VPH for gait improvement. Material and method: a randomized clinical trial was carried out with two intervention groups , applying it to one VPH group and the other ME.

The participants were residents of Geriatric Centers in the province of Seville, Spain with a score between 4 and 9 points according to the "Short Physical Performance Battery" scale (SPPB).

DETAILED DESCRIPTION:
This pilot study is a controlled and randomized clinical trial (simple ER) with two groups in parallel, comparing the combination of a multi-component therapeutic exercise protocol (ME) versus vestibular exercises (VPH) in over 70 years. The trial was approved by the Ethics Committee on Research with code 2410-N-19 and the study was conducted in accordance with the Helsinki Declaration.

ELIGIBILITY:
Inclusion Criteria:

* Males and females over 70 years of age.
* Subjects with a score between 4 and 9 points on the. "Short Physical Performance Battery"" (SPPB) scale

Exclusion Criteria:

* Patients unable to walk unaided or those who do not exceed the previous evaluation in SPPB.
* Polypharmacological patients (combined use of beta blockers, sulpiride or betahistin) were also excluded.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-04 (Actual); Primary Completion 2021-09-12 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Movement Capacity: SPPB (Short Physical Performance Battery) Physical Function Valuation Battery | Change from Baseline at 6 weeks
  The SPPB fitness rating battery consists of three parts: Balance rating, 4 metre gait assessment rating and the Time up and go test (TUG). From 0 (bad) to 12 (well) there is a score which describes de functionality
Speed test | Change from Baseline at 6 weeks
  Speed test. A participants walking speed over a 4 metre distance. This is a continuous quantitative variable measured in meters per second (m/s).
Test Time up and Go | Change from Baseline at 6 weeks
  The participants try to stand up and wlak 3 metres and return sitting. We must record the time.
  1) This is a continuous quantitative variable measured in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: MARINA LOPEZ LOPEZ-GARCIA, PT, Principal Investigator — University of Seville
Locations (1):
- Fundomar Elderly nursing home, Seville, Spain

IPD SHARING:
Plan to Share IPD: No
We are not to share de individual participants data to another investigators

REFERENCES:
- [Background] Iwasaki S, Yamasoba T. Dizziness and Imbalance in the Elderly: Age-related Decline in the Vestibular System. Aging Dis. 2014 Feb 9;6(1):38-47. doi: 10.14336/AD.2014.0128. eCollection 2015 Feb. PMID 25657851
- [Background] Agrawal Y, Carey JP, Della Santina CC, Schubert MC, Minor LB. Disorders of balance and vestibular function in US adults: data from the National Health and Nutrition Examination Survey, 2001-2004. Arch Intern Med. 2009 May 25;169(10):938-44. doi: 10.1001/archinternmed.2009.66. PMID 19468085
- [Background] Agrawal Y, Zuniga MG, Davalos-Bichara M, Schubert MC, Walston JD, Hughes J, Carey JP. Decline in semicircular canal and otolith function with age. Otol Neurotol. 2012 Jul;33(5):832-9. doi: 10.1097/MAO.0b013e3182545061. PMID 22699991
- [Background] Brown KE, Whitney SL, Marchetti GF, Wrisley DM, Furman JM. Physical therapy for central vestibular dysfunction. Arch Phys Med Rehabil. 2006 Jan;87(1):76-81. doi: 10.1016/j.apmr.2005.08.003. PMID 16401442
- [Background] Klatt BN, Ries JD, Dunlap PM, Whitney SL, Agrawal Y. Vestibular Physical Therapy in Individuals With Cognitive Impairment: A Theoretical Framework. J Neurol Phys Ther. 2019 Apr;43 Suppl 2(Suppl 2 Spec INTERNATIONAL CONFERENCE ON VESTIBULAR REHABILITATION):S14-S19. doi: 10.1097/NPT.0000000000000266. PMID 30883488
- [Background] Hall CD, Herdman SJ, Whitney SL, Cass SP, Clendaniel RA, Fife TD, Furman JM, Getchius TS, Goebel JA, Shepard NT, Woodhouse SN. Vestibular Rehabilitation for Peripheral Vestibular Hypofunction: An Evidence-Based Clinical Practice Guideline: FROM THE AMERICAN PHYSICAL THERAPY ASSOCIATION NEUROLOGY SECTION. J Neurol Phys Ther. 2016 Apr;40(2):124-55. doi: 10.1097/NPT.0000000000000120. PMID 26913496
- [Background] Swanenburg J, Wild K, Straumann D, de Bruin ED. Exergaming in a Moving Virtual World to Train Vestibular Functions and Gait; a Proof-of-Concept-Study With Older Adults. Front Physiol. 2018 Jul 31;9:988. doi: 10.3389/fphys.2018.00988. eCollection 2018. PMID 30108511
- [Background] Martins E Silva DC, Bastos VH, de Oliveira Sanchez M, Nunes MK, Orsini M, Ribeiro P, Velasques B, Teixeira SS. Effects of vestibular rehabilitation in the elderly: a systematic review. Aging Clin Exp Res. 2016 Aug;28(4):599-606. doi: 10.1007/s40520-015-0479-0. Epub 2015 Oct 28. PMID 26511625
- [Background] Baker MK, Atlantis E, Fiatarone Singh MA. Multi-modal exercise programs for older adults. Age Ageing. 2007 Jul;36(4):375-81. doi: 10.1093/ageing/afm054. Epub 2007 May 30. PMID 17537741
- [Background] Beato M, Dawson N, Svien L, Wharton T. Examining the Effects of an Otago-Based Home Exercise Program on Falls and Fall Risks in an Assisted Living Facility. J Geriatr Phys Ther. 2019 Oct/Dec;42(4):224-229. doi: 10.1519/JPT.0000000000000190. PMID 29698252
- [Background] Fishleder S, Petrescu-Prahova M, Harris JR, Leroux B, Bennett K, Helfrich CD, Kohn M, Hannon P. Predictors of Improvement in Physical Function in Older Adults in an Evidence-Based Physical Activity Program (EnhanceFitness). J Geriatr Phys Ther. 2019 Oct/Dec;42(4):230-242. doi: 10.1519/JPT.0000000000000202. PMID 29979352
- [Background] Canli S, Ozyurda F. A multi-modal exercise intervention that improves cognitive function and physical performance, elderly with mobility-related disability: a randomized controlled trial. J Sports Med Phys Fitness. 2020 Jul;60(7):1027-1033. doi: 10.23736/S0022-4707.20.10286-X. Epub 2020 Apr 6. PMID 32253894
- [Background] Gazzotti A, Meyer U, Freystaetter G, Palzer M, Theiler R, Abderhalden L, Bischoff-Ferrari HA. Physical performance among patients aged 70 + in acute care: a preliminar comparison between the Short Physical Performance Battery and the De Morton Mobility Index with regard to sensitivity to change and prediction of discharge destination. Aging Clin Exp Res. 2020 Apr;32(4):579-586. doi: 10.1007/s40520-019-01249-9. Epub 2019 Jul 8. PMID 31286430
- [Background] Casas-Herrero A, Anton-Rodrigo I, Zambom-Ferraresi F, Saez de Asteasu ML, Martinez-Velilla N, Elexpuru-Estomba J, Marin-Epelde I, Ramon-Espinoza F, Petidier-Torregrosa R, Sanchez-Sanchez JL, Ibanez B, Izquierdo M. Effect of a multicomponent exercise programme (VIVIFRAIL) on functional capacity in frail community elders with cognitive decline: study protocol for a randomized multicentre control trial. Trials. 2019 Jun 17;20(1):362. doi: 10.1186/s13063-019-3426-0. PMID 31208471
- [Background] Izquierdo M, Casas-Herrero A, Martinez-Velilla N, Alonso-Bouzon C, Rodriguez-Manas L; en representacion del Grupo de Investigadores. [An example of cooperation for implementing programs associated with the promotion of exercise in the frail elderly. European Erasmus + <<Vivifrail>> program]. Rev Esp Geriatr Gerontol. 2017 Mar-Apr;52(2):110-111. doi: 10.1016/j.regg.2016.03.004. Epub 2016 May 4. No abstract available. Spanish. PMID 27132063
- [Background] Rossi-Izquierdo M, Gayoso-Diz P, Santos-Perez S, Del-Rio-Valeiras M, Faraldo-Garcia A, Vaamonde-Sanchez-Andrade I, Lirola-Delgado A, Soto-Varela A. Prognostic factors that modify outcomes of vestibular rehabilitation in elderly patients with falls. Aging Clin Exp Res. 2020 Feb;32(2):223-228. doi: 10.1007/s40520-019-01185-8. Epub 2019 Apr 11. PMID 30977081
- [Background] Kundakci B, Sultana A, Taylor AJ, Alshehri MA. The effectiveness of exercise-based vestibular rehabilitation in adult patients with chronic dizziness: A systematic review. F1000Res. 2018 Mar 5;7:276. doi: 10.12688/f1000research.14089.1. eCollection 2018. PMID 29862019